CLINICAL TRIAL: NCT00958503
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Group Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of 14-Day Repeated-Dose Administration of Thiamphenicol (RUX 122) in Healthy Subjects
Brief Title: Effect of Thiamphenicol on EAAT2 and Other Biomarkers From Nasal Biopsied Tissue
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Psyadon Pharma (Industry)
Collaborators: SGS Life Sciences, a division of SGS Belgium NV (Other)
Responsible Party: Principal Investigator, Richard Chipkin, President and CEO, Psyadon Pharma
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EAAT2 Biomarker
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Healthy
Keywords: safety; biomarker; thiamphenicol; EAAT2
MeSH Terms: interventions — Thiamphenicol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Thiamphenicol (Active Comparator): Active comparator
  Interventions: Drug: Thiamphenicol

INTERVENTIONS:
Drug: Thiamphenicol — 750 and 1500 mg/day;tablets
  Other Names: Thiamphenicol, Urfamycine (trade name in Belgium)
  Arms: Thiamphenicol
Drug: Placebo — Matched tablets without active ingredient
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if two-weeks of dosing with thiamphenicol is safe and is able to change the levels of certain pre-specified biomarkers in nervous tissue taken from the nasal passages.

DETAILED DESCRIPTION:
Thiamphenicol has been proposed to increase the levels of the excitatory amino acid transporter 2 (EAAT2) in the nervous tissue. This study evaluated the ability of two weeks of treatment with thiamphenicol to increase EAAT2 in a nasal biopsy as a surrogate of brain nervous tissue.

ELIGIBILITY:
Inclusion Criteria:

* normal volunteers

Exclusion Criteria:

* less than 18 years
* older than 55 years

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-07; Primary Completion 2007-09 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Amount of EAAT2 RNA in nasal biopsy | Two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Chipokin, PhD, Principal Investigator — Ruxton Pharmaceuticals
Locations (1):
- SGS Research Unit - Stuivenberg, Antwerp, Belgium